CLINICAL TRIAL: NCT03740204
Title: The Role of Estrogen in the Neurobiology of Eating Disorders: A Study of Cognitive Flexibility and Reward in Eating Disorders
Brief Title: The Role of Estrogen in the Neurobiology of Eating Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Division Chief, Pediatric Endocrinology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH116205 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders; Hypoestrogenemia
Keywords: Adolescent; Amenorrhea; Anorexia Nervosa; Cognitive Flexibility; Dietary Restriction; Eating Disorders; Estrogen; Excessive Exercise; Females; Hypoestrogenemia; Reward
MeSH Terms: conditions — Feeding and Eating Disorders; Amenorrhea; Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 17-β estradiol with cyclic progesterone (Experimental)
  Interventions: Drug: 17-β estradiol transdermal patches with cyclic progesterone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo patch and pill

INTERVENTIONS:
Drug: 17-β estradiol transdermal patches with cyclic progesterone — 17-β estradiol transdermal patches (100 mcg 17-β estradiol/day) with cyclic progesterone (200 mg micronized progesterone daily for 12 days every month)
  Arms: 17-β estradiol with cyclic progesterone
Drug: Placebo patch and pill — Placebo patch and pill
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled study of the effects of transdermal estradiol versus placebo on cognitive flexibility, reward processing, and eating disorder pathology in hypoestrogenemic female adolescents and young adults (ages 14-35 years) with an eating disorder characterized by extreme dietary restriction and/or excessive exercise. Subjects will be randomized 1:1 to 12 weeks of transdermal estradiol with cyclic progesterone or placebo patches and cyclic placebo pills. Study visits include a screening visit to determine eligibility and visits at baseline, 8 weeks, and 12 weeks. Study procedures comprise behavioral, neuroimaging, and endocrine assessments.

ELIGIBILITY:
Inclusion criteria:

* Female
* 14-35 years
* Bone age ≥13.5 years (applicable only for participants <16 years)
* Clinically significant eating disorder characterized by restriction and/or excessive exercise and high drive for thinness
* Hypoestrogenemia: Oligo-amenorrhea defined as lack of menses for ≥3 months within a 6-month period of oligomenorrhea (cycle length ≥5 weeks) or absence of menses at >15 years if premenarchal or low estradiol levels evaluated by the study physician
* Low or normal weight defined by a body mass index that is <85th percentile for 14-18 year olds and a body mass index <25 kg/m2 for adults

Exclusion criteria:

* Suicidal ideation where outpatient treatment is determined unsafe by study clinician
* Other causes of oligo-amenorrhea, unless a study clinician determines that missed menstrual periods are more likely a consequence of restrictive eating
* Medications that contain estrogen ± progesterone within the past 3 months
* Levonorgestrel-releasing intrauterine device if subject is unable to provide two to three weekly blood samples for estradiol of if estradiol levels are determined to be too high by study doctor
* Neurological or psychiatric disorders that may impact neural circuitry of interest
* Lifetime history of seizure disorder or electroconvulsive therapy
* Pregnancy/breastfeeding
* Gastrointestinal tract surgery
* Contraindications to estrogen use
* Any other significant illness or condition that the investigator determines could interfere with study participation or safety or put the subject at any unnecessary risk

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in inhibition-switching performance on the Delis-Kaplan Executive Function System Color-Word Interference Test (D-KEFS CWIT) with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in Temporal Experience of Pleasure Scale (TEPS) Consummatory Pleasure score (Range: 8-48; direction: Higher values indicate more pronounced consummatory pleasure/better outcome) with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in delay discounting parameter k using the Monetary Choice Questionnaire with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in Eating Disorder Inventory-3 (EDI-3) Body Dissatisfaction score (Range: 0-36; direction: Higher values indicate more pronounced body dissatisfaction/worse outcome) with 17-β estradiol versus placebo | Baseline to 12 weeks
Change in EDI-3 Drive for Thinness score (Range: 0-28; direction: Higher values indicate more pronounced drive for thinness/worse outcome) with 17-β estradiol versus placebo | Baseline to 12 weeks

SECONDARY OUTCOMES:
Change in functional magnetic resonance imaging (fMRI) activation of the dorsolateral prefrontal cortex (DLPFC) and anterior cingulate cortex (ACC) during a task switching paradigm with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in fMRI activation of the ventromedial prefrontal cortex (VMPFC) and ventral striatum in response to reward receipt with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in fMRI activation of the VMPFC and ventral striatum during delay discounting with 17-β estradiol versus placebo | Baseline to 8 weeks
Change in the Eating Disorder Examination (EDE) Dietary Restraint subscale (Range: 0-6; direction: Higher values indicate more pronounced dietary restraint/worse outcome) with 17-β estradiol versus placebo | Baseline to 12 weeks
Change in caloric intake by 4-day food diary with 17-β estradiol versus placebo | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States